CLINICAL TRIAL: NCT05267236
Title: Impact Evaluation of the TYRO Couples Project
Brief Title: TYRO Couples Project Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: The RIDGE Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/34
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Couples

STUDY DESIGN:
Intervention Model Description: Treatment vs. Control Group Standard services delivered as primary services to participants in both study groups under a shared condition are: 20 hours of TYRO Dads curricula and 6 hours of Core Communication curricula. Optional services available to both study groups by selecting 1-3 hours of coursework from menu of courses that address a variety of needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-On Demand Format (Experimental): Treatment group participants receive TYRO Couples curriculum in an on-demand format that is delivered in five 2-hour weekly sessions for a total of 10 hours.
  Interventions: Other: Intervention #1: Treatment Group Receiving On-Demand TYRO Services
- Control-Virtual or In-Person Format (Experimental): Control group participants receive TYRO Couples curriculum in a live format (virtual or in-person) that is delivered in five 2-hour weekly sessions for a total of 10 hours.
  Interventions: Other: Intervention #2: Control Group Receiving In-Person TYRO Services

INTERVENTIONS:
Other: Intervention #1: Treatment Group Receiving On-Demand TYRO Services — Treatment group participants receive TYRO Couples curriculum in an on-demand format that is delivered in five 2-hour weekly sessions for a total of 10 hours.
  Arms: Treatment-On Demand Format
Other: Intervention #2: Control Group Receiving In-Person TYRO Services — Control group participants receive TYRO Couples curriculum in a live format (virtual or in-person) that is delivered in five 2-hour weekly sessions for a total of 10 hours.
  Arms: Control-Virtual or In-Person Format

SUMMARY:
This study uses an RCT design with repeated measures to test the impact of two different delivery formats for the TYRO Couples curriculum. Eligible study participants are males or females who are at least 18 years of age and within 9 months of release from incarceration. Incarcerated participants randomly assigned to the treatment group receive the TYRO Couples curriculum in-person, whereas those assigned to the comparison group experience an on-demand format. Study results that show no discernable differences in outcomes between groups will make it easier to serve more participants because service delivery formats can accommodate different life circumstances and preferences.

DETAILED DESCRIPTION:
The TYRO Couples curriculum Is based upon the Couples Communication curriculum, and was developed by a Christian, non-profit organization in Ohio called The RIDGE Project. The purpose of TYRO Couples is to provide training and opportunities for participants from families affected by the incarceration of a father to practice healthy relationship skills that build a foundation for healthy and successful marriages and lifelong partnerships. Curriculum components also address healthy financial and employment skills. Previous research suggests the TYRO Couples curriculum is efficacious in increasing skills related to: relationship building, couples communication, conflict resolution, and relationship satisfaction.

Typically, TYRO Couples is delivered in-person in a classroom setting. Using an in-person format results in a more personal, organic experience for participants but it requires a commitment that is difficult for some of them are unable to make because of the time and effort that is necessary to meet in a specific place for a predetermined amount of time. On-line access does not offer the same experience as in-person service delivery, but it does offer greater accessibility for participants to learn at their own pace in a self-directed learning environment of their own choosing. In theory, both formats offer program participants different types of access to service delivery and it is not clear if there is a disparate impact on the educational outcomes that define program benefits, which are improved attitudes, expectations and behaviors that promote healthy family relationships and economic stability for their households.

Testing the delivery format of TYRO Couples is important for several reasons. First, more research is needed to better understand which prison-based learning methods are more effective on marriage/intimate partner relationship and economic stability outcomes. Although there are some previous studies of best practices for prison-based learning, there are no studies, to our knowledge, that examine the effectiveness of on-demand learning on relationship and economic outcomes among couples affected by incarceration. Second, previous studies suggest that on-demand learning can be a helpful tool that empowers learners to digest the course material at their own pace. Learner control is a theory that derives from several motivational theory underpinnings, which includes attribution theory, motivation theory, and information processing theory. Previous research guided by learner control theory suggests that self-guided, on-demand learning is positively related to greater learner satisfaction and higher levels of learning compared with those who did not use this format.

Therefore, it is important that effective, prison-based learning methods are identified and used so that program participants can experience the most robust relationships and economic stability outcomes. Informed by the self-efficacy and learner control theory, the purpose of this study is to assess the extent to which TYRO Couples training delivered in an on-demand format has a disparate impact compared to in-person services on marriage/intimate partner relationships and economic stability outcomes among couples facing incarceration.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Adult (age 18 and older)
* Incarcerated
* Within 9 months of release in OH

Exclusion Criteria:

* Minor (under the age of 18)
* Not incarcerated
* Incarcerated but not within 9 months of release in OH

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- The RIDGE Project, McClure, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

REFERENCES:
- [Background] Allred, S. L., Harrison, L. D., & O'Connell, D. J. (2013). Self-Efficacy: An important aspect of prison-based learning. The Prison Journal, 93(2), 211 - 233. doi:10.1177/0032885512472964
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Chou, S., & Liu, C. (2005). Learning effectiveness in a web-based virtual learning environment: A learner-control perspective. Journal of Computer Assisted Learning, 21(1), 65 - 76.
- [Background] Cohen, J. 1988. Statistical Power Analysis for the Behavioral Sciences, 2nd Edition. Routledge.
- [Background] Foster, H., & Hagan, J. (2009). The Mass Incarceration of Parents in America: Issues of Race/ Ethnicity, Collateral Damage to Children, and Prisoner Reentry. The ANNALS of the American Academy of Political and Social Science, 623(1), 179-194. doi:10.1177/0002716208331123
- [Background] Frisco ML, Muller C, Frank K. Parents' Union Dissolution and Adolescents' School Performance: Comparing Methodological Approaches. J Marriage Fam. 2007 Aug 1;69(3):721-741. doi: 10.1111/j.1741-3737.2007.00402.x. PMID 20300482
- [Background] Johnson, B., Wubbenhorst, W., Schroeder, C., & Corcoran, K. E. (2014). Stronger Families, Stronger Society: An Analysis of the RIDGE Project, Inc. Baylor University. Waco, TX: Baylor Institute for Studies of Religion.
- [Background] La Vigne, N. G., Naser, R., Brooks, L. E., & Castro, J. L. (2005, November). Examining the effect of incarceration and in-prison. Journal of Contemporary Criminal Justice, 21(4), 314 - 335. doi:10.1177/1043986205281727
- [Background] Miller, S. L., Nunnally, E. W., & Wackman, D. B. (1976). A communication training program for couples. Social Casework, 57(1), 9 - 18.
- [Background] Manning WD. Cohabitation and Child Wellbeing. Future Child. 2015 Fall;25(2):51-66. doi: 10.1353/foc.2015.0012. PMID 26929590
- [Background] Shepherd, M. (2011). A statistical Analysis of Client Data from the Keeping Families and Inmates Together in Harmony (Keeping FAITH) Program for the RIDGE Project. Emporia, KS: Midwest Evaluation and Research.
- [Background] Siennick SE, Stewart EA, Staff J. EXPLAINING THE ASSOCIATION BETWEEN INCARCERATION AND DIVORCE. Criminology. 2014 Aug;52(3):371-398. doi: 10.1111/1745-9125.12040. PMID 25598544
- [Background] Visher, C. A., Debus-Sherrill, D., & Yahner, J. (2011). Employment after prison: A longitudinal study of former prisoners. Justice Quarterly, 28(5), 698 - 718. doi:10.1080/07418825.2010.535553
- [Background] Western B, Braga AA, Davis J, Sirois C. Stress and Hardship after Prison. AJS. 2015 Mar;120(5):1512-47. doi: 10.1086/681301. PMID 26421345
- [Background] Wildeman, C. (2014). How the criminal justice system shapes social inequality and the capacity of citizens: Parental Incarceration, child homelessness, and the invisible consequences of mass imprisonment. Annals of the American Academy of Political and Social Science, 651(1), 74-296.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from prisons within the Ohio Department of Rehabilitation and Corrections (ODRC).
  Enrollment took place between April 11, 2023, and continued through November 30, 2024
Pre-assignment Details: The only reason a participant would be excluded from the study after enrollment but before study assignment was if he/she did not provide consent to participate in the evaluation. Or, if he/she provided consent, then decided to revoke consent.
Period: Overall Study
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
Started | 403 | 417
Completed | 403 | 417
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format | Total
Number analyzed (Participants) | 403 | 417 | 820
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 403 | 415 | 818
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Full Range); unit: years] | 36 [19 to 65] | 36 [19 to 69] | 36 [19 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 43 | 61
  Male | 385 | 374 | 759
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 22 | 37
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 169 | 178 | 347
  White | 180 | 194 | 374
  More than one race | 11 | 8 | 19
  Unknown or Not Reported | 26 | 11 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 403 | 417 | 820

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure 1: Employment Attitudes
Description: What is the impact of on-demand delivery (treatment) compared to in-person delivery of the TYRO Couples curriculum (control) on employment attitudes six-months after enrollment?
  * 4 survey items independently measure the reported frequency of agreement with key co-parenting behaviors using categories on a 5-point scale (1 'Strongly Disagree', 2 'Disagree', 3 'Neither Agree nor Disagree', 4 'Agree', 5 'Strongly Agree').
  * Higher scores on 4 items indicate better outcomes (ex. - I can overcome almost any challenge to get a decent job.)
  Subscales were formed to add the four survey items together and were divided by four.
  The subscale ranges from 1-5 (the lowest someone can score is 1, the highest someone can score is 5-which is most favorable.
Time Frame: baseline to 6-month follow-up
Population: 111 participants completed the required survey items for this measure in the treatment group; 114 in the control group.
Measure: Mean (Standard Deviation); unit: score on subscale
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
Number analyzed (Participants) | 111 | 114
score on subscale | 4.16 (0.57) | 4.13 (0.59)

2. Primary Outcome: Primary Outcome Measure 2: Healthy Financial Attitudes
Description: What is the impact of on-demand delivery (treatment) compared to in-person delivery of the TYRO Couples curriculum (control) on financial attitudes six months after enrollment?
  * 3 survey items measure the reported agreement for key financial attitudes using categories on a 5-point employment attitudes scale (1 'Strongly Disagree', 2 'Disagree', 3 'Neither Agree Nor Disagree', 4 'Agree', 5 'Strongly Agree').
  * Higher scores on 3 items are negative (ex. - I am overwhelmed when I think about my financial situation.)
  Subscales were formed to add the three survey items together and were divided by three.
  The subscale ranges from 1-5 (the lowest someone can score is 1-which is most favorable, the highest someone can score is 5.
Time Frame: baseline to 6-month follow-up
Population: 114 participants in the treatment group responded to the survey items for this measure; 96 in the control group.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
Number analyzed (Participants) | 114 | 96
score on scale | 3.76 (0.63) | 3.78 (0.68)

3. Secondary Outcome: Secondary Outcome Measure 1: Partner Relationship Attitudes
Description: What is the impact of on-demand delivery (treatment) compared to in-person delivery of TYRO Couples curriculum (control) on partner relationship attitudes and expectations immediately after program completion?
  * 8 survey items measure the reported frequency of agreement with healthy partner relationship attitudes on a 5-point partner relationship attitudes scale (1 'Strongly Disagree', 2 'Disagree', 3 'Neither Agree Nor Disagree', 4 'Agree', 5 'Strongly Agree').
  * Higher scores on all items are positive (ex. - I want to grow old with my partner.)
  Subscales were formed to add the eight survey items together and were divided by eight.
  The subscale ranges from 1-5 (the lowest someone can score is 1, the highest someone can score is 5-which is most favorable).
Time Frame: baseline to immediately after program completion, up to 5 weeks
Population: 27 participants in the treatment group responded to the survey items for this measure; 25 in the control group.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
Number analyzed (Participants) | 27 | 25
score on scale | 4.35 (0.824) | 4.15 (1.113)

4. Secondary Outcome: Primary Outcome Measure 2: Relationship With Partner Behaviors
Description: What is the impact of on-demand delivery (treatment) compared to in-person delivery of the TYRO Couples curriculum (control) on partner relationship behaviors six months after enrollment?
  * 7 survey items measure the reported frequency the respondent engaged in a series of healthy behaviors with a partner using categories on a 7-point partner relationship behavior scale (1 'Never', 2 'Rarely', 3 'Sometimes', 4 'Often', 5 'Always').
  * Lower scores on all items are positive (ex. - How often do you and your partner disagree about religious matters?)
  Subscales were formed to add the seven survey items together and were divided by seven.
  The subscale ranges from 1-5 (the lowest someone can score is 1, the highest someone can score is 5-which is most favorable).
Time Frame: baseline to 6-month follow-up
Population: 44 participants in the treatment group responded to survey items in this measure; 47 in the control group. It was not required to be in a relationship to be in the study, so there was a very low completion rate for this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
Number analyzed (Participants) | 44 | 47
score on a scale | 3.39 (0.417) | 3.28 (0.471)

ADVERSE EVENTS:
Time Frame: six months through study completion
Description: The definition of adverse events does not differ from the clinicaltrials.gov definitions.
Arm/Group | Treatment-On Demand Format | Control-Virtual or In-Person Format
All-Cause Mortality (participants affected / at risk) | 0/820 | 0/820
Serious Adverse Events (participants affected / at risk) | 0/820 | 0/820
Other Adverse Events (participants affected / at risk) | 0/820 | 0/820

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT05267236/Prot_SAP_000.pdf